CLINICAL TRIAL: NCT06347731
Title: Varian ProBeam360° Proton Therapy System China Clinical Trial (Wuhan)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAR-2024-01
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Tumor, Solid
Keywords: Tumor; Radiation therapy; Proton therapy
MeSH Terms: conditions — Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Intervention Model Description: prospective, open-label, non-randomized, single-arm objective performance criteria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm objective performance criteria (OPC) (Other): According to the National Medical Products Administration (NMPA) Guidance on Proton and Carbon Ion treatment system clinical evaluation and clinical trial, The expected effective rate is 95%, and the target value is set at 80% of which the effective is defined as: tumor disease control rate = number of Complete Response (CR)+ Partial Response (PR)+ Stable Disease (SD)/the total number of subject*100%. Therefore, the clinical trial does not have a control group, but using single-arm objective performance criteria to evaluate ProBeam360 radiotherapy; the primary safety evaluation indicators is that CTCAE grade 3 toxic reaction ratio is lower than the acceptable value (5%), CTCAE grade 4 and 5 toxic reaction ratio is acceptable value (0%).
  Interventions: Device: Proton Radiation Therapy

INTERVENTIONS:
Device: Proton Radiation Therapy — All enrolled participants will be treated with Proton radiation therapy using the medical device Varian ProBeam360° Proton Therapy System. The screening period from informed consent to enrollment is expected to be 4 weeks, while the treatment period is 1 to 8 weeks. The period after the last treatment is divided into short-term follow-up which is 3 months after treatment completion and long-term follow-up which is 5 years after treatment completion.

SUMMARY:
This study is a clinical trial of prospective, single-center, single-arm objective performance criteria. This trial will be conducted with a total of 47 participants enrolled. All participants will be treated with radiation therapy using the medical device of Varian ProBeam360° Proton Therapy System (ProBeam360°), aim to compare the data with objective performance criteria (OPC) to evaluate the effectiveness and safety of ProBeam radiotherapy system for oncology patients, providing a clinical basis for the medical device registration.

DETAILED DESCRIPTION:
Tumors sites include Intracranial, head and neck, chest, abdomen, spine, pelvic cavity, extremity and other sites. The screening period from informed consent to enrollment is expected to be 4 weeks, while the treatment period is 1 to 8 weeks. The period after the last treatment is divided into short-term follow-up which is 3 months after treatment completion and long-term follow-up which is 5 years after treatment completion. The clinical trial with short-term follow-up fulfills the requirements for NMPA regulatory registration. All the end points claimed will be achieved in the short-term follow-up stage. The trial is defined as completion once short-term follow-up is finished.

And long-term follow-up report will be submitted for future post market evaluation when requested by NMPA.

ELIGIBILITY:
Inclusion Criteria (Major Criteria):

* Confirmed by cellular or histopathological diagnosis and/or evidence of imaging or laboratory tests, with a clinical diagnosis of benign, Patients with malignant intracranial tumors, as well as malignant solid tumors of the head and neck, chest, abdomen, spine, pelvis, and extremity;
* The target lesion is a measurable solid tumor, and the longest diameter of the lesion should be ≥10mm;
* Those who have an expected survival time of more than 6 months;
* Eastern Cooperative Oncology Group (ECOG) physical status is graded as 0~2;
* Females of childbearing potential with a negative blood or urine pregnancy test result within 7 days prior to the first treatment;

Exclusion Criteria (Major Criteria):

* Patients with contraindications to radiation therapy, including those with a known genetic predisposition to enhance the sensitivity of normal tissue radiotherapy or concomitant conditions leading to hypersensitivity to radiotherapy
* Patients with uncontrolled tumors other than the tumors to be treated, or patients with extensive metastases based on medical history or as judged by the investigator
* Proton radiation therapy area includes implanted pacemakers, defibrillators, cochlear implants, drug infusion pumps, other nerve stimulators, etc. (whether turned on or not); or passive implants that affect radiotherapy
* Tumor interventional treatment for the same lesion within 30 days prior to screening, such as transarterial chemoembolization (TACE), thermal ablation, etc.;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kunyu Yang, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from September 2024 to December 2024. The location of the study was in medical clinic.
Pre-assignment Details: Subjects meeting the inclusion/exclusion criteria and enrolled in the trial were treated with ProBeam360 Proton Therapy System (ProBeam360) unless the subject's status isn't fit for proton therapy prior to treatment during treatment planning and target area confirming. For example, if the subject's treatment plan indicated that within the target area wasn't suitable for radiation therapy, then should preclude from the trial.
Groups:
- single-arm objective performance criteria: The target value for efficiency should be at least 80%, with an expected 95%. Among them, the effective definition is CR+PR+SD (complete response CR, partial response PR, disease stable SD). The primary safety endpoints is that participants with Common Terminology Criteria for Adverse Events (CTCAE) grade 3 toxic reaction should be lower than 5%, CTCAE grade 4 and 5 toxic reaction rate is 0%. Therefore, the clinical trial did not have a control group, but using single-arm objective performance criteria.
  All enrolled subjects were treated with ProBeam Proton Therapy System. The period after the last treatment is divided into short-term follow-up and long-term follow-up, in which short-term follow-up is 3 months after treatment completion and long-term follow-up is 5 years after treatment completion. The clinical trial with short-term follow-up fulfills the requirements for NMPA regulatory registration. All the end points claimed will be achieved in the short-term follow-up stage. The trial is defined as completion once short-term follow-up finished.
  Long-term follow-up report will be submitted for future post market evaluation when requested by NMPA.
  Therefore, long-term follow-up result will not reported here.
Period: Overall Study
Arm/Group | single-arm objective performance criteria
Started | 47
Completed | 43
Not Completed | 4
Not completed — Death | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Single-arm Objective Performance Criteria: The target value for efficiency should be at least 80%, with an expected 95%. Among them, the effective definition is CR+PR+SD (complete response CR, partial response PR, disease stable SD). The primary safety endpoints is that participants with Common Terminology Criteria for Adverse Events (CTCAE) grade 3 toxic reaction should be lower than 5%, CTCAE grade 4 and 5 toxic reaction rate is 0%. Therefore, the clinical trial did not have a control group, but using single-arm objective performance criteria.
  All enrolled subjects were treated with ProBeam Proton Therapy System. The period after the last treatment is divided into short-term follow-up and long-term follow-up, in which short-term follow-up is 3 months after treatment completion and long-term follow-up is 5 years after treatment completion. The clinical trial with short-term follow-up fulfills the requirements for National Medical Products Administration (NMPA) regulatory registration. All the end points claimed will be achieved in the short-term follow-up stage. The trial is defined as completion once short-term follow-up finished.
  Long-term follow-up report will be submitted for future post market evaluation when requested by NMPA.
  Therefore, long-term follow-up result will not reported here.
Arm/Group | Single-arm Objective Performance Criteria
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (15.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 47

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness Measure: Tumor Disease Control Rate Reaches the Objective Performance Criteria (80%)
Description: At 3 months after the treatment completion, Disease control rate (DCR)will be assessed according to RECIST 1.1 criteria. DCR= The number of（complete response (CR)+partial response (PR)+stable disease (SD) ）/Total number of subject*100%.
  Tumor assessment measured by Magnetic Resonance Imaging (MRI)/Computed Tomography (CT) using Response Evaluation Criteria in Solid Tumors RECIST Version 1.1 (RECIST 1.1). CR, PR or SD were assessed through tumor size changes in CT or MRI images before and after treatment until 3-month follow-up visit.
  The target value for the main effectiveness evaluation (DCR) of the trial is 80% at 3 months after the end of the last radiotherapy session. If the lower limit of the 95% confidence interval of the experimental results is not less than 80%, then the DCR meets the trial Objective.
Time Frame: Primary effectiveness outcome measured change from baseline to 3 months ± 7 days after treatment completion
Measure: Count of Participants; unit: Participants
Groups:
- single-arm objective performance criteria (OPC): The target value for efficiency should be at least 80%, with an expected 95%. Among them, the effective definition is CR+PR+SD (complete response CR, partial response PR, disease stable SD). The primary safety endpoints is that participants with Common Terminology Criteria for Adverse Events (CTCAE) grade 3 toxic reaction should be lower than 5%, CTCAE grade 4 and 5 toxic reaction rate is 0%. Therefore, the clinical trial did not have a control group, but using single-arm objective performance criteria.
  All enrolled subjects were treated with ProBeam Proton Therapy System. The period after the last treatment is divided into short-term follow-up and long-term follow-up, in which short-term follow-up is 3 months after treatment completion and long-term follow-up is 5 years after treatment completion. The clinical trial with short-term follow-up fulfills the requirements for NMPA regulatory registration. All the end points claimed will be achieved in the short-term follow-up stage. The trial is defined as completion once short-term follow-up finished.
  Long-term follow-up report will be submitted for future post market evaluation when requested by NMPA.
  Therefore, long-term follow-up result will not reported here.
Arm/Group | single-arm objective performance criteria (OPC)
Number analyzed (Participants) | 43
Participants | 42

2. Primary Outcome: Percentage of Participants With Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 Toxic Reaction
Description: The percentage of participants with CTCAE grade 3 toxic reaction should be lower than 5%. Higher than 5% means worse outcome and will be considered as failure. AEs occurred in the clinical trial are recorded and scored by the investigator according to CTCAE version 5.0.
Time Frame: Primary safety outcome measured from enrollment to 3 months ± 7 days after treatment completion
Measure: Count of Participants; unit: Participants
Arm/Group | single-arm objective performance criteria
Number analyzed (Participants) | 47
Participants | 0

3. Primary Outcome: Percentage of Participants With Common Terminology Criteria for Adverse Events (CTCAE) Grade 4 and 5 Toxic Reaction
Description: The percentage of participants with toxic reaction of grade 4 and 5 should be 0%. If CTCAE grade 4 and 5 toxic reaction occured, It's not acceptable and the clinical trial is considered as failure.
  AEs occurred in the clinical trial are reported and scored by the investigator according to CTCAE version 5.0.
Time Frame: Primary safety outcome measured from enrollment to 3 months ± 7 days after treatment completion
Measure: Count of Participants; unit: Participants
Arm/Group | single-arm objective performance criteria
Number analyzed (Participants) | 47
Participants | 0

ADVERSE EVENTS:
Time Frame: The clinical trial started from participant enrollment to 3 months ± 7 days after the last treatment, up to 24 weeks. Long-term follow-up report (from 3-month follow-up till 5 years) will be submitted for future post market evaluation when requested by NMPA. Therefore, long-term follow-up result will not be reported here.
Arm/Group | single-arm objective performance criteria
All-Cause Mortality (participants affected / at risk) | 1/47
Serious Adverse Events (participants affected / at risk) | 6/47
Other Adverse Events (participants affected / at risk) | 40/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | single-arm objective performance criteria (N=47)
respiratory tract infection (Infections and infestations) | 2 (3)
Cerebral ischemic lesion (Nervous system disorders) | 2 (3)
Type 2 respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sudden death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | single-arm objective performance criteria (N=47)
Leukopenia (Investigations) | 7 (8)
neutropenia (Investigations) | 5 (7)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
renal insufficiency (Renal and urinary disorders) | 6 (6)
Elevated transaminase (Investigations) | 3 (3)
pulmonary infection (Infections and infestations) | 4 (4)
vomit (Gastrointestinal disorders) | 4 (4)
urinary tract infection (Infections and infestations) | 5 (5)
anemia (Blood and lymphatic system disorders) | 4 (4)
Weight loss (Metabolism and nutrition disorders) | 4 (4)
blood pressure elevation (Investigations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT06347731/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT06347731/SAP_001.pdf